CLINICAL TRIAL: NCT03903705
Title: A Phase Ib/II Study To Evaluate The Safety, Tolerability, Pharmacokinetic Profile And Preliminary Efficacy Of Fruquintinib Monotherapy Or Plus Sintilimab In Advanced Solid Tumors
Brief Title: : A Phase Ib/II Study To Evaluate Fruquintinib Monotherapy Or Plus Sintilimab In Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-013-00CH3
Record Dates: First submitted 2019-03-27; First posted 2019-04-04 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor
Keywords: Fruquintinib; Sintilimab; VEGFR; PD-1; Solid Tumor
MeSH Terms: interventions — HMPL-013; sintilimab

STUDY DESIGN:
Intervention Model Description: Open-Label Phase 1b/II Study of Fruquintinib in Combination with Sintilimab to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy in Patients with Advanced Solid Tumor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VEGFR cohort: (Experimental): Fruquintinib
  Interventions: Drug: Fruquintinib in Combination with Sintilimab

INTERVENTIONS:
Drug: Fruquintinib in Combination with Sintilimab — Fruquintinib plus Sintilimab:
  Cohort A: Fruquintinib 3 mg QD, oral dosing, 3 weeks on/1 weeks off +Sintilimab 200mg Q4W, intravenous dosing.
  Cohort B: Fruquintinib 4 mg QD, oral dosing, 3 weeks on/1 weeks off +Sintilimab 200mg Q4W, intravenous dosing
  Cohort C: Fruquintinib 5 mg QD, oral dosing, 2weeks on/1 weeks off + Sintilimab 200mg Q3W, intravenous dosing
  Cohort E: Fruquintinib 3 mg QD, continuous, oral dosing, + Sintilimab 200mg Q3W, intravenous dosing
  Fruquintinib monotherapy arm:
  Fruquintinib 5 mg QD, oral dosing, 3 weeks on/1 weeks off
  Patients will be treated until disease progression, death, unacceptable toxicity, loss of follow-up, withdrawal of consent or other conditions meet the end of treatment criteria.
  Other Names: Fruquintinib

SUMMARY:
This is a phase Ib/II study to evaluate the safety, tolerability, PK profile and preliminary efficacy of fruquintinib monotherapy or plus sintilimab for advanced solid tumors. This study includes fruquintinib plus sintilimab treatment arm (dose escalation phase and dose expansion phase), and fruquintinib monotherapy arm.

DETAILED DESCRIPTION:
This study is composed of Fruquintinib plus sintilimab treatment arm and Fruquintinib monotherapy arm.

Fruquintinib plus sintilimab treatment arm:

* Dose escalation phase: it is planned to enroll about 26-39 patients
* Dose expansion phase: it is planned to enroll about 309-329 patients, including about 140 patients with endometrial cancer

Fruquintinib monotherapy arm: about 13 patients with advanced endometrial cancer

ELIGIBILITY:
Inclusion Criteria:

* Have fully understood and voluntarily sign the ICF for this study (the icf must be signed before any trial-specific procedures are performed);
* Age of 18-75 years (inclusive); BMI ≥18.5 kg/m2;
* Tumor types:
* Fruquintinib plus sintilimab treatment arm
* Dose escalation phase: patients with histologically or cytologically confirmed inoperable or metastatic advanced solid tumors (including but not limited to HCC, ovarian cancer, endometrial cancer, thymic cancer, NSCLC, renal cell carcinoma);
* Dose expansion phase: histologically or cytologically confirmed inoperable metastatic advanced HCC (Barcelona Clinic Liver Cancer [BCLC] stage B or C), advanced renal cell carcinoma with clear cell component, advanced endometrial cancer, advanced gastric adenocarcinoma or gastroesophageal junction adenocarcinoma, advanced colorectal adenocarcinoma, advanced NSCLC, advanced cervical cancer, etc.;
* Fruquintinib monotherapy treatment arm: histologically or cytologically confirmed metastatic advanced endometrial cancer that cannot be surgically resected or treated with radical radiotherapy;
* In the expansion phase, patients should agree to provide tissue specimens for detection of PD-L1 expression levels and/or MSI or dMMR status;
* Requirement for prior systemic antitumor therapy:
* Fruquintinib plus sintilimab treatment arm:
* Dose escalation phase: patients who have failed standard treatment (PD or intolerable toxicity after treatment), have no available standard treatment or cannot receive standard treatment (such as economic limitations);
* Dose expansion phase:
* Part 1
* Patients (HCC, renal cell carcinoma, endometrial cancer, gastric adenocarcinoma or gastroesophageal junction adenocarcinoma, colorectal adenocarcinoma, cervical cancer, NSCLC) should have PD or intolerable toxicity after 1 standard treatment, or cannot receive standard treatment (such as economic limitations or patient's wishes, etc.). Among them, requirements of standard treatment are defined as follows:
* Patients with HCC who have received 1 molecular targeted therapy (sorafenib or lenvatinib) or/and systemic chemotherapy (arsenious acid monotherapy or oxaliplatin-based combination therapy);
* Patients with renal cell carcinoma who have received 1 standard systemic antitumor therapy (sunitinib, sorafenib, pazopanib, axitinib, cabozantinib, bevacizumab plus IFN-α, temsirolimus);
* Patients with endometrial cancer who have received ≤2 line of platinum-based double drug systemic antitumor therapy (excluding hormonal therapy) and had PD or Grade ≥3 SAE, or had recurrence or PD after completion of at least 4 cycles of platinum-based double drug chemotherapy. Patients with recurrence or metastasis during or within 12 months after completion of neoadjuvant/adjuvant chemotherapy with platinum-based regimen are considered to have received first-line treatment (4 cycles are required for neoadjuvant/adjuvant chemotherapy, and if less than 4 cycles, it is also eligible to have PD or Grade ≥3 SAE during the treatment);
* Patients with cervical cancers who have recurrent or metastasized squamous cell carcinoma, adenocarcinoma, or adeno-squamous carcinoma after at least one line of platinum-based chemotherapy (patients are considered to have received first-line treatment if they have recurrent or metastasized during or within 6 months after platinum-based neoadjuvant or adjuvant chemotherapy);
* Patients with gastric adenocarcinoma and gastroesophageal junction adenocarcinoma who have failed prior standard chemotherapy and can provide tumor tissues for PD-L1 expression detection with CPS ≥1;
* Patients with colorectal adenocarcinoma previously treated with fluoropyrimidine+leucovorin calcium+platinum or irinotecan+cetuximab/bevacizumab.
* Advanced NSCLC (stage IV NSCLC diagnosed per AJCC 8th version):
* Patients with negative driver gene (EGFR/ALK/ROS-1 negative) who have failed prior standard treatment or have intolerable toxicity, or cannot receive or are unwilling to receive current standard treatment, and with PD-L1 expression level TPS (tumor proportion score) ≥1% tested by central laboratory arranged by the sponsor.
* Patients with NSCLC diagnosed with squamous cell carcinoma do not require test of EGFR mutation, ALK and ROS1 fusion per current diagnosis and treatment guidelines. Other non-squamous NSCLC patients can be included if they have a prior test report demonstrating no driver gene mutation/rearrangement (EGFR, ALK, ROS1); if there is no prior corresponding gene report, archived or fresh tissue needs to be collected for testing at the study site, or at the central laboratory arranged by sponsor.
* Patients who have recurrence or metastasis during or within 6 months after prior neoadjuvant/adjuvant therapy are considered as having received first-line therapy.
* Part 2
* To enroll patients with renal cell carcinoma who have not received systemic therapy, the specific requirements are as follows:
* Patients with renal cell carcinoma have not received any prior systemic antitumor therapy for renal cell carcinoma (patients with recurrence or PD >6 months after postoperative adjuvant chemotherapy can be enrolled), and patients with prior cytokine therapy are allowed.
* Fruquintinib monotherapy arm: patients with histologically or cytologically confirmed advanced recurrent or metastatic endometrial cancer who cannot be surgically resected or treated with radical radiotherapy and have failed at least 1 standard treatment (including PD and intolerable toxicity).
* ECOG performance status (ECOG PS) of 0 or 1;
* Child-Pugh Class A (<7 points) for liver function, only applicable to patients with HCC;
* Measurable tumor lesions per RECIST 1.1, where patients with gastric tumor are required to have measurable lesions outside of the stomach (in the dose escalation phase, patients with only the evaluable lesions are acceptable); if the lesion priorly treated with local therapy (radiotherapy, ablation, interventional therapy, etc.) is the only lesion, there must be definite imaging evidence of PD for that lesion;
* Laboratory test results of bone marrow, liver and kidney function, and coagulation function within 7 days before the first dose should meet the following criteria (no blood transfusion, blood products, granulocyte colony-stimulating factor or other hematopoietic stimulating factor correction within 7 days before the laboratory test)

  * Absolute neutrophil count (ANC) ≥1.5×109/L and platelets ≥100×109/L (platelets ≥80×109/L in patients with HCC) and hemoglobin ≥90 g/L;
  * Serum total bilirubin (TBIL) ≤1.5 times upper limit of normal (×ULN);
  * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤1.5×ULN without liver metastases; ALT and/or AST ≤3×ULN with liver metastases and HCC;
  * Serum albumin ≥28 g/L;
  * Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min (calculated per Cockcroft-Gault formula);
  * Protein urine < 2+; if protein urine ≥ 2+, 24-hour protein urine quantification should be <1 g;
  * International normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5×ULN (except for prophylactic use of anticoagulant drugs);
* Life expectancy of ≥12 weeks;
* Female of childbearing potential must have a negative blood pregnancy test within 7 days before the first dose. Male or female patients of childbearing potential should voluntarily use an effective contraceptive method during the study and within 6 months after the last dose of study drug, such as double-barrier contraceptive method, condom, oral or injectable contraceptives, intrauterine device, abstinence, etc. All female patients are considered to be of childbearing potential unless they are postmenopausal, have undergone artificial menopause, or are sterilized (hysterectomy, excision of both adnexa).

Exclusion Criteria:

* The AEs related to prior antitumor therapy which do not recover to ≤ CTCAE Grade 1 before the first dose, except alopecia and peripheral neurotoxicity of CTCAE Grade ≤2 caused by platinum chemotherapy;
* Patients with other malignant tumors (except cured cutaneous basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ) within 5 years before screening, only applicable to patients in expansion phase;
* Histological diagnosed fibrolamellar HCC, sarcomatoid HCC or mixed components of the above pathological types; or gastric squamous cell carcinoma or gastric adenosquamous carcinoma; or carcinosarcoma or sarcoma (endometrial cancer); or pathological diagnosis MSI-H or dMMR (endometrial cancer)
* Patients with previous or screening stage central nervous system (CNS) metastasis during screen period (for lung cancer patients with brain metastasis who have prior treatment, if there is no evidence of radiographic progression within ≥4 weeks before the first dose of study drug, and are clinically stable for ≥2 weeks after treatment, and have discontinued corticosteroids within 3 days before the first dose, the patient could be enrolled; for patients with untreated, asymptomatic lung cancer with brain metastasis [i.e., no neurological symptoms, no need for corticosteroid or antiepileptic treatment, no brain metastasis >1.5 cm in long diameter, no significant edema around brain metastasis], they could be enrolled);
* Systemic antitumor therapy approved or under study within 4 weeks before the first dose, including but not limited to: chemotherapy (oral fluoropyrimidines washout period of 2 weeks), endocrine therapy, biological immunotherapy, targeted therapy (small molecule targeted therapy washout period of 2 weeks or 5 half-lives, whichever shorter), Traditional Chinese Medicine treatment (Traditional Chinese Medicine treatment with definite antitumor indications in the instructions, a 1-week washout period before the first dose is acceptable);
* Radical radiotherapy (including more than 25% bone marrow radiotherapy) within 4 weeks before the first dose;
* Brachytherapy (such as implantation of radioactive particles) within 60 days before the first dose;
* Patients previously treated with any anti-programmed cell death receptor 1 (PD-1) antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibody (or any other antibody acting on T cell costimulation or checkpoint pathway) (only for the fruquintinib plus sintilimab treatment arm), or fruquintinib;
* Corticosteroids (dose >10 mg/day prednisone or equivalent of other corticosteroids) or other immunosuppressive drugs for systemic treatment within 4 weeks before the first dose; nasal spray, inhalation or other topical use of corticosteroids (i.e., no more than 10 mg/day prednisone or equivalent of other glucocorticoids) are allowed;
* Patients with any active autoimmune disease requiring systemic treatment (i.e., use of disease remission drugs, glucocorticoids or immunosuppressive drugs) within the past 2 years; patients who only need replacement therapy (thyroid, adrenal or pituitary dysfunction with thyroid, insulin or physiological glucocorticoid replacement therapy) can be enrolled;
* Any live or attenuated live vaccines within 4 weeks before the first dose or planned administration during the study;
* Major surgical operation within 60 days before the first dose;
* Any surgery or invasive treatment within 4 weeks before the first dose (stable fistula formation required for fistulization for 4 weeks, except needle biopsy, venous fistula); or unhealed wounds, ulcers, fractures;
* Uncontrolled malignant pleural effusion, ascites or pericardial effusion (defined as not effectively controlled by diuretics or paracentesis, as judged by the investigator);
* Patients with hypertension uncontrolled by drugs, defined as: systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg;
* Patients with any disease or condition that affects drug absorption, or the patient could not take the drug orally;
* Strong cytochrome P450 (CYP) 3A4 inducer/inhibitor, p-glycoprotein (P-gp) substrate and breast cancer resistance protein (BCRP) substrate within 2 weeks or less than 5 half-lives (whichever is longer) before the first dose;
* Patients with active gastric and duodenal ulcer, ulcerative colitis and other gastrointestinal diseases or unresected tumor with active bleeding, or other conditions that may cause gastrointestinal bleeding and perforation as judged by the investigator; or patients with prior gastrointestinal perforation or gastrointestinal fistula who had not recovered after surgical treatment;
* Patients with evidence or history of bleeding tendency (such as melena, hematemesis, hemoptysis, bloody feces, etc.) within 2 months before the first dose, regardless of severity;
* Tumor invading major vascular structures, such as pulmonary artery, superior/inferior vena cava, etc. found during screening, with greater risk of bleeding judged by the investigator;
* Patients with a history of arterial thrombosis or deep venous thrombosis within 6 months before the first dose; or patients with stroke events and/or transient ischemic attack within 12 months; except that patients with thrombosis caused by implantable venous infusion pump or catheter, or patients with stable superficial venous thrombosis after conventional anticoagulant therapy;
* Patients with clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina or coronary artery bypass grafting within 6 months before the first dose; congestive heart failure of New York Heart Association (NYHA) class ≥ 2; left ventricular ejection fraction (LVEF) of < 50%;
* Patients with an active infection or unexplained fever (body temperature >38.5oC) during the screening period or before the first dose;
* Patients with active pulmonary tuberculosis who are receiving anti-tuberculosis treatment or received anti-tuberculosis treatment within 1 year before the first dose;
* Patients with prior and current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired pulmonary function and other conditions that may interfere with the detection and treatment of suspected drug-related pulmonary toxicity;
* Known human immunodeficiency virus (HIV) infection;
* Known history of clinically significant liver disease, including active viral hepatitis, (hepatitis B virus surface antigen [HBsAg] and/or hepatitis B virus core antibody [HbcAb] positive, hepatitis B virus [HBV] DNA >10000 copies/mL or > 2000 IU/mL; hepatitis C virus [HCV] antibody positive and HCV RNA positive), or other active hepatitis, clinically significant moderate to severe cirrhosis;
* Other clinical drug treatment that has not been approved or marketed in China within 4 weeks before the first dose;
* Women who are pregnant (positive pregnancy test before dose) or breastfeeding;
* Known hypersensitivity to any component of the sintilimab, fruquintinib formulation, or prior history of severe allergy to any other monoclonal antibody;
* Patient with any other condition or laboratory abnormalities that, in the opinion of the investigator, will increase the risk of study participation or interfere with the interpretation of study results, and is not suitable for the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Dose escalation phase: Safety outcome evaluation - DLT, MTD/RP2D | From first dose to 30 days post the last dose
  Dose escalation phase: To evaluate the safety and tolerability of fruquintinib plus sintilimab for advanced solid tumors in the dose escalation phase, to observe dose-limiting toxicity (DLT), the maximum tolerated dose (MTD) and/or to determine the recommended phase 2 dose (RP2D) and administration strategy of the combination therapy.
Dose expansion phase (except EMC cohort): efficacy outcome evaluation - ORR based on the investigator's tumor assessment | very 6 weeks since Cycle1 Day 1, and every 12 weeks after Week 48, until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent
  Dose expansion phase (except endometrial cancer [EMC] cohort): ORR assessed by investigator
Dose expansion phase (EMC cohort): efficacy outcome evaluation - ORR based on IRC's tumor assessment | Every 6 weeks since Cycle1 Day 1, and every 12 weeks after Week 48, until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent
  Dose expansion phase (EMC cohort): ORR by IRC
Fruquintinib monotherapy arm: efficacy outcome evaluation - ORR based on investigator's tumor assessment | Every 6 weeks since Cycle1 Day 1, and every 12 weeks after Week 48, until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent
  Fruquintinib monotherapy arm: ORR by investigator

SECONDARY OUTCOMES:
Immunogenicity Assessments for Anti-drug Antibody(ADA) | From Cycle 1, 2, 4, 6, 8, 12 (each cycle is 28 days) and the safety visit for Sintilimab until disease progression or death or new anti-cancer therapy or withdrawal of consent
  Immunogenicity Assessments for Anti-drug Antibody(ADA)
pharmacokinetics (PK) Assessments | From Cycle 1 for Fruquintinib; Cycle 1, 2, 3, 4 for Sintilimab in the dose escalation phase, and Cycle 1, 2, 4, 12 for dose expansion phase.
  To evaluate the PK profile of fruquintinib plus sintilimab
Dose expansion phase (except EMC cohort): Efficacy outcome evaluation - DCR, PFS, OS, DoR, TTR based on the investigator's tumor assessment | Every 6 weeks since Cycle1 Day 1, and every 12 weeks after Week 48, until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent
  Dose expansion phase (except EMC cohort): DCR, PFS, OS, DoR, TTR by investigator
Dose expansion phase (EMC cohort): Efficacy outcome evaluation - ORR, DCR, PFS, OS, DoR, TTR based on the investigator's tumor assessment | Every 6 weeks since Cycle1 Day 1, and every 12 weeks after Week 48, until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent
  Dose expansion phase (EMC cohort): ORR, DCR, PFS, OS, DoR, TTR by investigator
Dose expansion phase (EMC cohort): Efficacy outcome evaluation - DCR, PFS, OS, DoR, TTR based on the IRC's tumor assessment | Every 6 weeks since Cycle1 Day 1, and every 12 weeks after Week 48, until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent
  Dose expansion phase (EMC cohort): DCR, PFS, OS, DoR, TTR by IRC
Safety outcome evaluation | From first dose to 30 days post the last dose
  Overall incidence of AEs, incidence of Grade ≥ 3 AEs, etc.
Biomarker evaluation | From first dose to 30 days post the last dose
  Detect the expression of PD-L1 and/or other biomarkers in tumor tissues of patients, and analyze the relevant efficacy to provide reference for determining the dominant population.

OTHER OUTCOMES:
Exploratory outcome | From first dose to 30 days post the last dose
  Evaluate the potential biomarkers related to the antitumor effect of fruquintinib plus sintilimab.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu X, Wang J, Wang D, Li G, Zhang J, Chen H, Yang H, Zhou Q, Wang K, Wu Y, Yi T, Liu J, Huang Y, Bai Y, Wang K, Jiang K, Lou H, An R, Li X, Pan Y, Wang Y, Tao W, Song K, Kang Y, Li Y, Shi W, Liu A, Yang Y, Wang Y, Chen K, Shi H, Lu P, Tan P, Fan S, Shi M, Su W. Fruquintinib plus sintilimab in patients with advanced endometrial cancer with mismatch-repair proficient status: a multicenter, single-arm, phase Ib/II trial. Nat Commun. 2025 Dec 21;17(1):658. doi: 10.1038/s41467-025-67375-3. PMID 41423492
- [Derived] Xu H, Yao X, He Z, Luo H, Li G, Guo J, Diao L, Fan Y, Li Y, Fan J, Hu X, Lu P, Shi H, Chen K, Tan P, Fan S, Shi M, Su W, Ye D. Fruquintinib Plus Sintilimab in Patients with Treatment-Naive and Previously Treated Advanced Renal Cell Carcinoma: Results from a Phase Ib/II Clinical Trial. Target Oncol. 2025 Jan;20(1):113-125. doi: 10.1007/s11523-024-01120-6. Epub 2025 Jan 13. PMID 39806128
- [Derived] Guo Y, Zhang W, Ying J, Zhang Y, Pan Y, Qiu W, Fan Q, Xu Q, Ma Y, Wang G, Guo J, Su W, Fan S, Tan P, Wang Y, Luo Y, Zhou H, Li J. Phase 1b/2 trial of fruquintinib plus sintilimab in treating advanced solid tumours: The dose-escalation and metastatic colorectal cancer cohort in the dose-expansion phases. Eur J Cancer. 2023 Mar;181:26-37. doi: 10.1016/j.ejca.2022.12.004. Epub 2022 Dec 13. PMID 36628898